CLINICAL TRIAL: NCT05074329
Title: Multi-center, Prospective, Randomized, Controlled, Clinical Trial for Idiopathic Hip Pain Using Peripheral Nerve Stimulation
Brief Title: Clinical Trial for Idiopathic Hip Pain Using Peripheral Nerve Stimulation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Uro Medical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TWIST 31-00105
Record Dates: First submitted 2021-09-29; First posted 2021-10-12 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2021-09

CONDITIONS: Idiopathic Hip Pain; Chronic Hip Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Active (Active Comparator): Subjects randomized to the Active group, programming parameters will be set, and therapy will be delivered for a minimum of 2-hours per day for the duration of the study.
  Interventions: Device: Moventis PNS
- Delayed (Placebo Comparator): The delayed group will begin 2-hour stimulation/day at the 3-Month visit.
  Interventions: Device: Moventis PNS

INTERVENTIONS:
Device: Moventis PNS — Moventis PNS is indicated for pain management in adults who have severe intractable chronic pain of peripheral nerve origin.

SUMMARY:
This is a prospective, randomized, multi-center study in which 300 evaluable subjects will be randomized 1:1 to receive Active or Delayed therapy with Moventis PNS. Subjects in the Delayed group will start with therapy at 3-month visit follow up.

DETAILED DESCRIPTION:
This is a prospective, randomized, controlled, multi-center study in which 300 evaluable subjects will receive Moventis PNS. Target subjects will have idiopathic hip pain.

Subjects will be randomized into either a delayed or immediate continuation group. Devices will be activated post-op in accordance to the randomization assignment. Subjects randomized to the Active group, programming parameters will be set, and therapy will be delivered for a minimum of 2-hours per day for the duration of the study. Implanted subjects will be educated on the use of the transmitter. Programming changes can be done as needed during this time period to maximize clinical response according to pre-programmed settings. Subjects randomized to the Delayed group will begin 2-hour stimulation/day at the 3-Month visit.

The primary endpoint is to demonstrate clinically significant improvements in the pain of patients in the active group compared to the subjects in the delayed group. The primary endpoint is defined as >50% pain relief at 3-months as measured by the Visual Analog Scale (VAS) without increase in baseline pain medications. Improvement will be assessed in relation to the clinical outcome measures of pain, with a target of >50% pain relief.

ELIGIBILITY:
Inclusion Criteria:

* Capable of giving informed consent;
* Capable and willing to follow all study related procedures;
* Women and men >18 years of age;
* Diagnosis of hip pain;
* Baseline VAS score of >5;
* >50% temporary relief from temporary nerve diagnostic evaluation;
* No evidence of anatomic abnormalities that could jeopardize device placement;
* Able to operate programmer, recharger, study assessments and provide accurate responses;
* Appropriate candidate for the implant procedure.

Exclusion Criteria:

* An active implantable electronic device regardless of whether stimulation is ON or OFF;
* Pregnant or plan to become pregnant during study;
* Less than 1-year post-partum and/or are breast-feeding;
* Symptoms existing for less than 6 months;
* Multiple complaints that will not be amenable to study;
* Current diagnosis of a Neurological disease;
* Daily opioid usage exceeding CDC recommendations;
* Dependency on utilizing wearable or transcutaneous monitoring device (hearing aids, continuous glucose monitors, etc.);
* Conditions requiring recurring MRI evaluation or diathermy procedures;
* Uncontrolled diabetes (HbA1C > 8.5);
* Known or suspected substance abuse within the last 2-years;
* Uncontrolled major depression or uncontrolled psychiatric disorders;
* Worker's compensation claimants;
* History of adverse reaction to local anesthetic drugs;
* History of coagulopathy or bleeding disorder;
* Anatomical restrictions such that device placement is not possible;
* Chronic or acute conditions that could interfere with the interpretations of the outcome assessment for pain and bodily function;
* Have a life expectancy of less than 1-year;
* Neurogenic or vascular claudication;
* Inability to achieve appropriate positioning and inability to understand informed consent and protocol;
* Deemed unsuitable for enrollment by investigator based on history or physical examination.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2021-11 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Rate of Change in Pain Relief: >50% pain relief as measured by Visual Analog Scale | 3 Months
  Improvement pain defined as a >50% pain relief as measured by VAS without increase in baseline medications. To demonstrate clinically significant improvements in the pain of subjects in the active group compared to the subjects in the delayed group.
Adverse Events | 3 Months
  Device- and procedure-related Adverse Events (AE) rate at 3-months.

SECONDARY OUTCOMES:
Change in Hip Pain: measured by Hip Pain Questionnaire | 3, 6, 9, 12, 24, 36-months
  Current hip pain will be accessed and the history of hip pain will be recorded.
Rate of Change in Pain Relief: >50% pain relief as measured by Visual Analog Scale | 6, 9, 12, 24, 36-Months
  Improvement pain defined as a >50% pain relief as measured by VAS without increase in baseline medications. To demonstrate clinically significant improvements in the pain of subjects in the active group compared to the subjects in the delayed group.

IPD SHARING:
Plan to Share IPD: Yes
Upon study completion